CLINICAL TRIAL: NCT02577510
Title: A Comparison Between Ultrasound- and Neurostimulation-Guided Lateral Femoral Cutaneous Nerve Block
Brief Title: Comparing Ways to Freeze the Nerve That Provides Thigh Sensation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Canadian Forces Health Services Centre Ottawa (Other)
Responsible Party: Principal Investigator, Gaurav Gupta, MD FRCPC, Canadian Forces Health Services Centre Ottawa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: #2014-005-
Record Dates: First submitted 2015-10-14; First posted 2015-10-16 (Estimated); Results first posted 2017-09-15 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Meralgia Paresthetica
Keywords: Lateral Femoral Cutaneous Nerve Block; Meralgia Parasthetica; nerve stimulator; ultrasound
MeSH Terms: conditions — Femoral Neuropathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nerve Stimulation- Xylocaine injection (Experimental): Anesthesia of the lateral femoral cutaneous nerve using local anesthetic will be randomly assigned on the right or left side to receive nerve stimulation-xylocaine or ultrasound guided -xylocaine injections in all patients. One patient will therefore have both nerve stimulation AND ultrasound guided injections, only the side of the injection will be randomly assigned to one of the two modalities. Once one technique has been used to freeze one side, the other side will be frozen using the other technique.
  Interventions: Drug: Nerve Injection- Nerve Stimulator
- Ultrasound guided Xylocaine injection (Experimental): Anesthesia of the lateral femoral cutaneous nerve using local anesthetic will be randomly assigned on the right or left side to receive nerve stimulation-xylocaine or ultrasound guided -xylocaine injections in all patients. One patient will therefore have both nerve stimulation AND ultrasound guided injections, only the side of the injection will be randomly assigned to one of the two modalities. Once one technique has been used to freeze one side, the other side will be frozen using the other technique.
  Interventions: Drug: Nerve Injection - Ultrasound

INTERVENTIONS:
Drug: Nerve Injection- Nerve Stimulator — For the neurostimulation nerve injection technique, the initial puncture site will be located medial to the anterosuperior iliac spine, just caudal to the inguinal ligament [7]. The 22-gauge insulated needle will be connected to a stimulator set at a current of 1.5 mA, a pulse width of 300 ms and a frequency of 2 Hz. A paresthesia referred to the lateral aspect of the thigh at a minimal stimulatory threshold of 0.6 mA (0.3ms) will be sought prior to the injection of local anesthetic [7]. A total of 5cc of 2%Xylocaine will be injected for the nerve injection/anesthesia.
  Other Names: Lateral Femoral Cutaneous Nerve Block- Neurostimulation
  Arms: Nerve Stimulation- Xylocaine injection
Drug: Nerve Injection - Ultrasound — For the ultrasound nerve injection group, after skin disinfection, the inguinal region of patients will be scanned using a high-frequency (6 to 13 MHz) linear array transducer covered with a sterile plastic cover. An ultrasound image showing the inguinal ligament and anterior superior iliac spine (ASIS) will be obtained. Using an out-of-plane technique, a 22-gauge nerve block needle will be inserted 1-2 cm medial to ASIS. The needle will be advanced until its tip rests under the inguinal ligament, immediately ventral to the iliopsoas muscle [6]. A total of 5cc of 2%Xylocaine will be injected for the nerve injection/anesthesia.
  Other Names: Lateral Femoral Cutaneous Nerve Block- Ultrasound
  Arms: Ultrasound guided Xylocaine injection

SUMMARY:
Background

The sensation on the outside of portion of our thighs is provided by a nerve called the lateral femoral cutaneous nerve (LFCN). The investigators can inject freezing around the nerve to reduce the feeling around the thigh (i.e. anesthesia). Anesthesia, or freezing, of the lateral femoral cutaneous nerve can reduce pain for patients having A) hip and knee surgery [1,2], B) removal of a skin graft [3], and C) wound care. In addition, damage to the LFCN (i.e. Meralgia Paresthetica) has been associated with body armour and gun belt use in military and police personnel [4]. Although generally a benign condition, compression or injury to this nerve can be painful and require treatment. In addition, the actual variability in sensory distribution for this nerve has not been elucidated in a topographical fashion and will be measured in this study.

Finding the most efficient and effective method for anesthesia of the LFCN can improve and positively impact the quality of pain control for patients. Ultrasound has improved the accuracy and efficiency of various other regional anesthesia techniques, and could also impact the safety. Therefore the investigators hypothesize that ultrasound guided lateral femoral cutaneous nerve block using the subinguinal technique will be statistically more efficacious and efficient when compare to neurostimulation based blockade.

DETAILED DESCRIPTION:
Purpose of the Study:

The goal of this study is to compare the ultrasound-guided subinguinal injection technique to the neurostimulation-guided injection technique for lateral femoral cutaneous nerve block. The neurostimulation technique uses an electrical field to stimulate the nerve when a needle is close proximity. One older study showed it is better than using landmarks in achieving anesthesia of the lateral femoral cutaneous nerve, but no studies have compared it to using ultrasound to freeze the nerve [7]. The primary outcome will be relative efficiency, i.e. the total anesthesia-related time (defined as the sum of performance and onset times). This is looking at how long it takes for the procedure (needle insertion, medication injection), plus the time it takes for the thigh to go numb. Secondary outcomes will include relative success rate, procedural discomfort, number of needle passes and topographical sensory distribution of this nerve in this cohort of patients .

Methodology:

Selection of Human Subjects:

With the approval of the Defence Research & Development Canada Human Research Ethics Committee (HREC), a total of 27 volunteers will be recruited. Subjects will be recruited by advertising within the CF Health Services Centre Facility and by email notification to CF members in the National Capital region through the DWAN. If there is insufficient volunteers, those people that have volunteered, will be contacted by email to inquire if they are aware of any other people that maybe be interested in volunteering so that the study can be finalized. If they know if anyone, they will be asked to forward the initial email to those people, asking them to contact the investigator if they wish to have more information. Interested civilian volunteers and Class "A" reservists will be approached from the cohort of patients that responded to the original communication email.

Once patients have submitted their names for consideration, they will be contacted to review whether they meet inclusion/exclusion criteria.

Data Analyses:

the investigators expect the success rates to be similar for both groups. However our hypothesis is that the performance time and the onset time could be different. Therefore the main outcome is the total anesthesia-related time (sum of performance and onset times). According to Shannon et al [7], the total anesthesia-related time for the neurostimulation technique is 10.1 +/- 4.7 min (performance time: 9.5 +/- 4.7 min and onset time: 0.8 +/- 0.9 min). Using a paired T-test to compare both techniques, a difference of 30% in total anesthesia time would represent an effect size of 0.74 and require a total of 17 subjects undergoing bilateral blocks to obtain a 2-tailed α error of 0.05 and a ß error of 0.2. Since onset and total anesthesia-related times can only be measured for successful blocks and since the investigators expect a success rate of 85% for neurostimulation, the investigators will recruit 25 patients to account for those who do not reach the postulated end point.

Normality of the continuous data will first be assessed with the Kolmogorov-Smirnov test. Continuous data will then analyzed using a paired T-test. For categorical data, the Mann-Whitney U test and Chi-square test will be used as appropriate. Hypotheses tested will be 2-tailed. P < 0.05 will be considered statistically significant.

Risks:

Participation in this study will be voluntary and volunteers can withdraw consent at any time without having any effect on access to future medical care. There will likely minor discomfort during the procedure similar to having freezing before a dental procedure or blood drawn. Patients can ask us to stop the procedure at any time. The chance of minor discomfort for up to a day or two after the injection can occur and can be managed with over the counter acetaminophen or ibuprofen. The investigators do not expect any limitations to daily activities.

Furthermore, side effects associated with lateral femoral cutaneous nerve blocks have not been reported and are likely rare. [8].

Confidentiality/Anonymity

Patients' confidentiality/anonymity will be protected through two mechanisms:

* research subjects are identified by serial numbers
* access to patient's research data will be restricted to primary investigators only

Approximate Time Involvement

The approximate time commitment is 1.5 hour.

Roles and Responsibilities of Research Team

Recruitment, study planning and organization will be done by Gaurav Gupta. Technical procedures, data collection and manuscript preparation will be shared tasks by the entire research team.

ELIGIBILITY:
Inclusion Criteria:

* male and female between 18 and 60 years old
* American Society of Anesthesiologists classification 1-3

Exclusion Criteria:

* adults who are unable to give their own consent
* pre-existing neuropathy (assessed by history and physical examination) -
* coagulopathy (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. platelets ≤ 100, International Normalized Ratio ≥ 1.4 or prothrombin time ≥ 50)
* renal failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. creatinine ≥ 100)
* hepatic failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. transaminases ≥ 100)
* allergy to local anesthetic agents local anesthetic
* pregnancy based on patient self report of last menstrual cycle. If a patient wish/insist on participating in the study, and pregnancy status is unclear, a urine pregnancy test will be offered. Also risk of Lidocaine in pregnancy will be discussed with the patient as currently classified. We will convey that this risk is currently classified as a Risk Class B, which means that animal-reproduction studies have not demonstrated a fetal risk but there are no controlled studies in pregnant women. We will also discuss that animal-reproduction studies have shown an decrease in maternal fertility), but that was not confirmed in controlled studies in women in the first trimester and there is no evidence of a risk in later trimesters,
* prior surgery in the hip and lateral leg region
* prior lumbar surgery
* previous pelvic fracture
* previous L1, L2 or L3 lumbar radiculopathy, plexopathy or meralgia paresthetica
* chronic pain syndromes requiring opioid intake

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2015-11; Primary Completion 2016-02 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav Gupta, MD, Principal Investigator — CF Health Centre Ottawa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim JH, Cho MR, Kim SO, Kim JE, Lee DK, Roh WS. A comparison of femoral/sciatic nerve block with lateral femoral cutaneous nerve block and combined spinal epidural anesthesia for total knee replacement arthroplasty. Korean J Anesthesiol. 2012 May;62(5):448-53. doi: 10.4097/kjae.2012.62.5.448. Epub 2012 May 24. PMID 22679542
- [Background] Capdevila X, Biboulet P, Bouregba M, Rubenovitch J, Jaber S. Bilateral continuous 3-in-1 nerve blockade for postoperative pain relief after bilateral femoral shaft surgery. J Clin Anesth. 1998 Nov;10(7):606-9. doi: 10.1016/s0952-8180(98)00097-x. PMID 9805704
- [Background] Shteynberg A, Riina LH, Glickman LT, Meringolo JN, Simpson RL. Ultrasound guided lateral femoral cutaneous nerve (LFCN) block: safe and simple anesthesia for harvesting skin grafts. Burns. 2013 Feb;39(1):146-9. doi: 10.1016/j.burns.2012.02.015. Epub 2012 May 30. PMID 22657583
- [Background] Fargo MV, Konitzer LN. Meralgia paresthetica due to body armor wear in U.S. soldiers serving in Iraq: a case report and review of the literature. Mil Med. 2007 Jun;172(6):663-5. doi: 10.7205/milmed.172.6.663. PMID 17615854
- [Background] Fowler IM, Tucker AA, Mendez RJ. Treatment of meralgia paresthetica with ultrasound-guided pulsed radiofrequency ablation of the lateral femoral cutaneous nerve. Pain Pract. 2012 Jun;12(5):394-8. doi: 10.1111/j.1533-2500.2011.00522.x. Epub 2011 Dec 7. PMID 22151457
- [Background] Hara K, Sakura S, Shido A. Ultrasound-guided lateral femoral cutaneous nerve block: comparison of two techniques. Anaesth Intensive Care. 2011 Jan;39(1):69-72. doi: 10.1177/0310057X1103900111. PMID 21375093
- [Background] Shannon J, Lang SA, Yip RW, Gerard M. Lateral femoral cutaneous nerve block revisited. A nerve stimulator technique. Reg Anesth. 1995 Mar-Apr;20(2):100-4. PMID 7605755
- [Background] Stan TC, Krantz MA, Solomon DL, Poulos JG, Chaouki K. The incidence of neurovascular complications following axillary brachial plexus block using a transarterial approach. A prospective study of 1,000 consecutive patients. Reg Anesth. 1995 Nov-Dec;20(6):486-92. PMID 8608066
- [Background] Corujo A, Franco CD, Williams JM. The sensory territory of the lateral cutaneous nerve of the thigh as determined by anatomic dissections and ultrasound-guided blocks. Reg Anesth Pain Med. 2012 Sep-Oct;37(5):561-4. doi: 10.1097/AAP.0b013e318261c8b6. PMID 22878522

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We enrolled 21 participants and randomized the sides for each modality.
Units Other Than Participants: sides
Groups:
- Nerve Stimulation- Xylocaine Injection: Anesthesia of the lateral femoral cutaneous nerve using local anesthetic will be randomly assigned on the right or left side to receive nerve stimulation-xylocaine or ultrasound guided -xylocaine injections in all patients. One patient will therefore have both nerve stimulation AND ultrasound guided injections, only the side of the injection will be randomly assigned to one of the two modalities. Once one technique has been used to freeze one side, the other side will be frozen using the other technique.
  Nerve Injection- Nerve Stimulator: For the neurostimulation nerve injection technique, the initial puncture site will be located medial to the anterosuperior iliac spine, just caudal to the inguinal ligament [7]. The 22-gauge insulated needle will be connected to a stimulator set at a current of 1.5 mA, a pulse width of 300 ms and a frequency of 2 Hz. A paresthesia referred to the lateral aspect of the thigh at a minimal stimulatory threshold of 0.6 mA (0.3ms) will be sought prior
- Ultrasound Guided Xylocaine Injection: Nerve Injection - Ultrasound: For the ultrasound nerve injection group, after skin disinfection, the inguinal region of patients will be scanned using a high-frequency (6 to 13 MHz) linear array transducer covered with a sterile plastic cover. An ultrasound image showing the inguinal ligament and anterior superior iliac spine (ASIS) will be obtained. Using an out-of-plane technique, a 22-gauge nerve block needle will be inserted 1-2 cm medial to ASIS. The needle will be advanced unt
Period: Overall Study
Arm/Group | Nerve Stimulation- Xylocaine Injection | Ultrasound Guided Xylocaine Injection
Started | 21; 21 sides | 21; 21 sides
Completed | 21; 21 sides | 21; 21 sides
Not Completed | 0; 0 sides | 0; 0 sides

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 17
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 21
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.7 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: Anesthesia Related Time
Description: The main outcome will be the total anesthesia-related time, defined as the sum of performance and onset times
Time Frame: less than 30 minutes
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: sides
Arm/Group | Nerve Stimulation | Ultrasound
Number analyzed (Participants) | 21 | 21
Number analyzed (sides) | 21 | 21
seconds | 554 (366.9) | 480 (251.9)
Statistical Analysis 1: Comparison: Nerve Stimulation vs Ultrasound; Statistical analysis was performed using SPSS Version 21 statistical software (IBM, Armonk, New York). For continuous data, normality was fi rst assessed with the Lilliefors test and then analyzed using a paired t test. Data that did not have a normal distribution, as well as ordinal data, was analyzed using Wilcoxon's signed ranks or McNemar's test. All P values presented were 2-sided and values inferior to 0.05 were considered signifi cant; Test type: Other; p = 0.05, t-test, 1 sided

2. Secondary Outcome: Success Rate
Description: percentage of patients with successful block
Time Frame: less than 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Nerve Stimulation | Ultrasound
Number analyzed (Participants) | 21 | 21
Participants | 16 | 20

3. Secondary Outcome: Needle Pass
Description: how often needle changes angle to make target
Time Frame: less than 30 minutes
Measure: Mean (Standard Deviation); unit: attempts
Units Other Than Participants: sides
Arm/Group | Nerve | Ultrasound
Number analyzed (Participants) | 21 | 21
Number analyzed (sides) | 21 | 21
attempts | 9.5 (12.2) | 3.2 (2.9)

4. Secondary Outcome: Pain With Procedure
Description: visual analogue scale- 0-10 - 0 is equal to no pain, while 10 is equal to maximum pain
Time Frame: less than 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: sides
Arm/Group | Nerve Stimulation- Xylocaine Injection | Ultrasound Guided Xylocaine Injection
Number analyzed (Participants) | 21 | 21
Number analyzed (sides) | 21 | 21
units on a scale | 4.0 (2.2) | 4.6 (2.2)

ADVERSE EVENTS:
Time Frame: within 30 minutes post injection and 72 hours of injection
Groups:
- Ultrasound Guided Xylocaine Injection; Nerve Stimulation Guided Xylocaine Injection: Adverse event collected for this side with this intervention.
Arm/Group | Ultrasound Guided Xylocaine Injection | Nerve Stimulation Guided Xylocaine Injection
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 1/21 | 0/21
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ultrasound Guided Xylocaine Injection (N=21) | Nerve Stimulation Guided Xylocaine Injection (N=21)
Femoral Block (Nervous system disorders) | 1 (1) | 0 (0) — femoral nerve block

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No